CLINICAL TRIAL: NCT02080169
Title: Safety and Efficacy of Combined Sedation With Midazolam and Dexmedetomidine in ICU Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Qilu Hospital of Shandong University (Other)
Collaborators: Chinese Medical Association (Network)
Responsible Party: Principal Investigator, Qian Zhai, Intensive Care Unit, Qilu Hospital of Shandong University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CMAqiluICU
Record Dates: First submitted 2014-02-25; First posted 2014-03-06 (Estimated); Last update posted 2014-03-06 (Estimated); Status verified 2014-03

CONDITIONS: Delirium
Keywords: Intensive care unit; Mechanical ventilation; Combined sedation
MeSH Terms: conditions — Delirium | interventions — Midazolam; Dexmedetomidine; Fentanyl

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- midazolam (Experimental): Initiative dosage of midazolam is 0.05 mg/kg given intravenously, the maintenance dosage is 0.01-0.05 mg/kg/h, drug dosage is adjusted by target sedation level.
  Interventions: Drug: midazolam; Drug: Fentanyl
- Dexmedetomidine (Experimental): The loading dose of dexmedetomidine is 0.5-0.8 μg/kg given intravenously more than 10 min, the maintenance dosage is 0.2-0.7 μg/kg/h,the drug dosage is adjusted by target sedation level.
  Interventions: Drug: Dexmedetomidine; Drug: Fentanyl
- midazolam & dexmedetomidine (Experimental): Initiative dosage of midazolam is 0.05 mg/kg given intravenously, The loading dose of dexmedetomidine is 0.5-0.8 μg/kg given intravenously more than 10 min(given or not according to patients' condition),.
  The maintenance dosage of midazolam is 0.01-0.05 mg/kg/h, the maintenance dosage of dexmedetomidine is 0.2-0.7 μg/kg/h,the drug dosage is adjusted by target sedation level.
  Interventions: Drug: midazolam; Drug: Dexmedetomidine; Drug: Fentanyl

INTERVENTIONS:
Drug: midazolam — If the target sedation level is not obtained using the above recommended dosage, midazolam 0.01-0.05 mg/kg is added every 10-15min, until the target sedation level is obtained.
  If it is over sedation (RASS -3 to -5), and reduction of the dosage of the sedation drug could not ease the situation, and then stop the sedation until the target sedation level is obtained.
  Other Names: Liyuxi
  Arms: midazolam; midazolam & dexmedetomidine
Drug: Dexmedetomidine — If the target sedation level is not obtained using the above recommended dosage, midazolam 0.01-0.05 mg/kg is added every 10-15min, until the target sedation level is obtained.
  If it is over sedation (RASS -3 to -5), and reduction of the dosage of the sedation drug could not ease the situation, and then stop the sedation until the target sedation level is obtained.
  Other Names: Yisi
  Arms: Dexmedetomidine; midazolam & dexmedetomidine
Drug: Fentanyl — Fentanyl is used as analgesic drug in order to obtain the VAS <3.

SUMMARY:
It is well known that ICU patients need sedation. Now no ideal sedation drug existed and every sedation drug has its advantage and disadvantage,so combined sedation may use the advantage and avoid the disadvantage of the sedation drug according to the patients'condition. Until now, there is rare study about the combined sedation or sequenced sedation of different sedation drug.The purpose of the study is to explore the value of combined sedation with midazolam and dexmedetomidine compared to single drug sedation in ICU, so as to seek an ideal sedation protocol that could reduce the cost of treatment,obtain the appropriate sedation not under sedation or over sedation,reduce the incidence of delirium, reduce the adverse event of sedation.

ELIGIBILITY:
Inclusion Criteria:

1. ICU patients needing sedation
2. 18 years or older
3. mechanically ventilated for less than 96 hours prior to start of study drug.

Exclusion Criteria:

1. Trauma and burn patients as admitting diagnosis.
2. Dialysis of all types.
3. Pregnant or lactation.
4. Neuromuscular blockade other than for intubation.
5. Epidural or spinal analgesia.
6. General anesthesia prior to or planned after the start of study drug infusion
7. Serious central nervous system pathology(acute stroke, uncontrolled seizures,severe dementia).
8. Acute hepatitis or severe liver disease (Child-Pugh class C).
9. Unstable angina or acute myocardial infarction.
10. Left ventricular ejection fraction less than 30%,heart rate less than 50/min. 11.Second or third degree heart block.

12.Allergy to the study drug. 13.Systolic blood pressure less than 90 mm Hg despite continuous infusions of 2 vasopressors before the start of study drug infusion.

14. Patients with renal insufficiency were randomized and treated; however, patients were discontinued if they required dialysis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2014-02; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
The total time within target sedation level | From sedation drug is used to weaning from sedation up to 28 days.
  1. Sedation level with RASS score is recorded every 4 hours during sedation.
  2. When target sedation was not obtained, sedation drug dosage changed and when adverse event needed to be treated, the sedation level is also recorded.
  3. The adjustment of sedation drug is recorded.

SECONDARY OUTCOMES:
The dosage of sedation/analgesic drug | From sedation/analgesic drug is used to weaning from sedation/analgesic up to 28 days.
  Record the induced and maintained dosage of sedation/opioid analgesic drug. The total dosage of sedation/opioid analgesic drug. The added dosage of midazolam.
Duration of mechanical ventilation | From beginning to weaning from ventilation up to 28 days..
  The duration of mechanical ventilation is recorded.
Economic outcome | From admitted to ICU until ventilation and sedation stopped and participants discharged from ICU up to 28 days.
  The cost of sedation drug used is recorded. The cost of mechanical ventilation is recorded. The cost of ICU residency is recorded.
Satisfactory of patients to ICU stay from admitted until discharged from ICU | Assessed at time of 1 week participants discharged from ICU.
  Evaluated the satisfactory of patients to ICU. Using scores including 0 to 10. 0 presents extremely dissatisfied and 10 presents extremely satisfied.
Delirium | From sedation drug is used to weaning from sedation, up to 28 days.
  Delirium is evaluated when daily sedation interruption is done during sedation. Delirium incidence is recorded using CAM-ICU. Treatment of delirium is recorded including drug,dosage and method of administration.
Vital signs | From sedation drug is used to weaning from sedation, up to 28 days.
  Heart rate(HR),main arterial pressure(MAP),respiratory rate(RR),pulse saturate of oxygen(SPO2) are recorded every 4 hours. When sedation drug dosage changed and adverse events treated,the vital signs is also recorded.
  Gas blood analysis index is recorded when the daily interruption is done and when the SPO2 is less 90% or 10% decrease than normal.
Duration of ICU stay | From date of admission until participants discharged from ICU up to 28 days.
  Record when participants discharged form ICU.

CONTACTS AND LOCATIONS:
Overall Officials: Da W Wu, Doctor., Study Director — Qilu Hospital of Shandong University
Locations (1):
- Department ICU, Shandong university affiliated Qilu Hospital., Jinan, Shandong, China